CLINICAL TRIAL: NCT00001277
Title: Studies of Hyperparathyroidism and Related Disorders
Brief Title: Studies of Elevated Parathyroid Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 910085; 91-DK-0085 (Other: NIH Clinical Center)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-02-07

CONDITIONS: Hyperparathyroidism; Hypercalcemia; Parathyroid Neoplasm; Multiple Endocrine Neoplasia; MEN1
Keywords: Hypoglycemia; Genetics; Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism; Hypercalcemia; Parathyroid Neoplasms; Multiple Endocrine Neoplasia; Hypoglycemia | interventions — gallium Ga 68 dotatate; fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary hyperparathyroidism (No Intervention): Patients with confirmed or suspected primary hyperparathyroidism or complications
- DOTATATE and F-DOPA (Experimental): Patients scanned using imaging agents 68GALLIUM-DOTATATE and 18F-DOPA
  Interventions: Drug: 68Ga-Dotatate; Drug: 18F-DOPA

INTERVENTIONS:
Drug: 68Ga-Dotatate — 68Ga-Dotatate PET/CT will be administered prior to a PET/CT scan to detect known and occult primary and metastatic bronchial, gastrointestinal and pancreatic neuroendocrine tumors.
  Arms: DOTATATE and F-DOPA
Drug: 18F-DOPA — 18F-DOPA PET/CT will be administered prior to a whole-body scan to detect known and occult primary and metastatic bronchial, gastrointestinal and pancreatic neuroendocrine tumors.
  Arms: DOTATATE and F-DOPA

SUMMARY:
Observational Phase: Patients whose parathyroid activity is elevated above normal are referred to as having hyperparathyroidism. This study will help researchers better understand the causes of hyperparathyroidism and to evaluate and improve methods for diagnosis and treatment. Patients diagnosed with or suspected of having hyperparathyroidism will be selected to participate. In addition, patients with related conditions, such as parathyroid tumors, will also be selected.

Subjects will be asked to provide blood and urine for testing to confirm their condition. They will then be surgically treated by removal of the parathyroid gland(s) (parathyroidectomy). Subjects with parathyroid tumors will undergo several diagnostic tests to determine the exact location of the tumor as well as the tumor's activity. The tests may include; ultrasounds, nuclear scanning, CT scans, MRI, and specialized blood testing.

Sometimes parathyroidectomy leads to hypoparathyroidism. Options for treating the patients after the surgical procedure will also be addressed. Calcium and Vitamin D supplements are typically the mainstay of post parathyroidectomy therapy. Other potential treatments include transplanting the parathyroid gland(s) to other areas of the body.

Clinical Trial: An imaging substudy was added to this protocol in 2018. Patients with multiple endocrine neoplasia type 1 (MEN1) will have 68Gallium-Dotatate Positron Emission Tomography (PET) - Computed Tomography (CT), 18F-DOPA PET/CT, MRI, and CT scans and the number of lesions detected by each of these types of scans will be compared.

DETAILED DESCRIPTION:
Observational: Patients with confirmed or suspected primary hyperparathyroidism or complications therefrom (such as postoperative hypoparathyroidism) will be admitted for diagnosis and treatment. The principal diagnostic components are calcium in serum and urine, parathyroid hormone in serum, and mutation tests on germline or tumor DNA. Patients with moderate to severe primary hyperparathyroidism will be treated. Treatment will be mainly by parathyroidectomy. Other options are medications or no intervention. Patients with a hyperparathyroid syndrome may be managed for their extraparathyroid features. Preoperative testing to localize parathyroid neoplasm(s) will be used usually and with more extended methods in cases with prior neck surgery. Preoperative tumor localization tests will be selected according to clinical indications from the following: ultrasound, technetium-thallium scan, computerized tomography, magnetic resonance imaging, fine needle aspiration for parathyroid hormone assay, selective arteriogram, selective venous catheterization for parathyroid hormone assay. Options for management of postoperative hypocalcemia include calcium, vitamin D analogs, parathyroid autografts and synthetic parathyroid hormone. Research specimens may consist of blood or tumors.

Clinical Trial: An imaging substudy was added to this protocol in 2018. Patients with MEN1 will have 68Ga-Dotatate PET/CT, 18F-DOPA PET/CT, MRI, and CT scans and the number of lesions detected by each of these types of scans will be compared.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients who have genetically confirmed MEN1 or clinical criteria of MEN1.
* For females: Negative urine pregnancy test OR post-menopausal for at least 2 years OR patient has had a hysterectomy

EXCLUSION CRITERIA:

* Serious underlying medical conditions that restrict diagnostic testing or therapy such as renal failure or congestive cardiac failure
* Patients unable or unwilling to give informed consent
* Pregnant or lactating women: Pregnant women are excluded from this study because the effects of 68Ga-DOTATATE in pregnancy are not known. Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of 68Ga-DOTATATE in the mother, women who are breastfeeding are also excluded from this study
* Patients that have recognized concurrent active infection
* Patients with known hypersensitivity to carbidopa, or who are concurrently taking a nonselective monoamine oxidase (MAO) inhibitor..

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1553 (Actual)
Dates: Start 1993-12-15 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smita Jha, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1991-DK-0085.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Hyperparathyroidism - Incomplete Data: Patients with confirmed or suspected primary hyperparathyroidism or complications who are missing age and other baseline data because of changes in data management system
Period: Overall Study
Arm/Group | Primary Hyperparathyroidism - Incomplete Data | Primary Hyperparathyroidism | DOTATATE and F-DOPA
Started | 634 | 900 | 19
Completed | 634 | 900 | 16
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — The tracer F-DOPA did not meet Quality Control Standards | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Age is not available for 634 participants in the primary hyperparathyroidism arm because the necessary records are not in the current computer system
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Hyperparathyroidism - Incomplete Data | Primary Hyperparathyroidism | DOTATATE and F-DOPA | Total
Number analyzed (Participants) | 634 | 900 | 19 | 1553
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — Population: These data are not available because of changes to the data management system. Most were enrolled before the year 2000.
  Years
    number analyzed (Participants) | 0 | 900 | 19 | 919
    (all) |  | 48 [36 to 60] | 54 [38 to 64] | 48 [36 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 409 | 582 | 6 | 997
  Male | 225 | 318 | 13 | 556
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 0 | 14 | 14
  Unknown or Not Reported | 634 | 900 | 4 | 1538
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 0 | 4
  Asian | 0 | 25 | 0 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 100 | 1 | 101
  White | 0 | 719 | 16 | 735
  More than one race | 0 | 13 | 0 | 13
  Unknown or Not Reported | 634 | 38 | 2 | 674
Region of Enrollment [Number; unit: participants]
  United States | 634 | 900 | 19 | 1553

OUTCOME MEASURES:

1. Primary Outcome: Type of Hyperparathyroidism
Description: The purpose of this study is to understand the causes of primary hyperparathyroidism, to evaluate and improve methods for diagnosis and treatment, and to provide insight into the mechanisms of normal parathyroid function. Hereditary causes of primary hyperparathyroidism will be characterized. Patients were categorized as follows:
  1. MEN1: Diagnosed by demonstration of a germline variant in MEN1 gene or one of the following: a) two of three primary MEN1 manifestations b) one primary MEN1 manifestation with a family member with MEN1.
  2. Other familial: Non-MEN1 patients who had a positive family history of hyperparathyroidism suspicious for underlying germline predisposition syndrome.
  3. Sporadic: Patients who did not have a positive family history of hyperparathyroidism.
  4. Unknown: No data to help categorize the patients in any of the above categories.
Time Frame: First year
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Hyperparathyroidism - Incomplete Data | Primary Hyperparathyroidism | DOTATATE and F-DOPA
Number analyzed (Participants) | 634 | 900 | 19
Participants
  MEN1 | 90 | 276 | 19
  Other familial | 61 | 116 | 0
  Sporadic | 456 | 419 | 0
  Unknown - insufficient information | 27 | 89 | 0

2. Primary Outcome: Organs With Identified Lesions
Description: For each organ, agreement between 68Ga-DOTATATE and 18F-DOPA
Time Frame: Days 1-6
Population: Imaging was only conducted in the "DOTATATE and F-DOPA" Arm/Group and therefore results are only reported for this arm
Measure: Count of Participants; unit: Participants
Groups:
- DOTATATE and F-DOPA: Patients who received both DOTATATE and F-DOPA scans
Arm/Group | DOTATATE and F-DOPA
Number analyzed (Participants) | 16
Participants
  All locations: No lesions by Dotatate or F-DOPA | 1
  All locations: Lesions by F-DOPA only | 0
  All locations: Lesions by Dotatate only | 7
  All locations: Lesions by Both | 8
  Lung: No lesions by Dotatate or F-DOPA | 13
  Lung: Lesions by F-DOPA only | 0
  Lung: Lesions by Dotatate only | 0
  Lung: Lesions by Both | 3
  Gastrointestinal: No lesions by Dotatate or F-DOPA | 12
  Gastrointestinal: Lesions by F-DOPA only | 0
  Gastrointestinal: Lesions by Dotatate only | 3
  Gastrointestinal: Lesions by Both | 1
  Pancreas: No lesions by Dotatate or F-DOPA | 3
  Pancreas: Lesions by F-DOPA only | 0
  Pancreas: Lesions by Dotatate only | 9
  Pancreas: Lesions by Both | 4
  Duodenum: No lesions by Dotatate or F-DOPA | 9
  Duodenum: Lesions by F-DOPA only | 0
  Duodenum: Lesions by Dotatate only | 6
  Duodenum: Lesions by Both | 1
  Liver: No lesions by Dotatate or F-DOPA | 11
  Liver: Lesions by F-DOPA only | 0
  Liver: Lesions by Dotatate only | 3
  Liver: Lesions by Both | 2
  Adrenal: No lesions by Dotatate or F-DOPA | 12
  Adrenal: Lesions by F-DOPA only | 1
  Adrenal: Lesions by Dotatate only | 3
  Adrenal: Lesions by Both | 0
  Lymph nodes: No lesions by Dotatate or F-DOPA | 7
  Lymph nodes: Lesions by F-DOPA only | 0
  Lymph nodes: Lesions by Dotatate only | 4
  Lymph nodes: Lesions by Both | 5

3. Primary Outcome: Number of Lesions Identified
Description: The total number of lesions identified by each imaging modality
Time Frame: Days 1-6
Population: Imaging was only conducted in the "DOTATATE and F-DOPA" Arm/Group and therefore results are only reported for this arm. This outcome is only reported for the 16 patients who had both scans
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | DOTATATE and F-DOPA
Number analyzed (Participants) | 16
Number analyzed (Lesions) | 134
Lesions
  No lesions by Dotatate or F-DOPA | 44
  Lesions by F-DOPA only | 1
  Lesions by Dotatate only | 67
  Lesions by Both | 22

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Primary Hyperparathyroidism - Incomplete Data | Primary Hyperparathyroidism | DOTATATE and F-DOPA
All-Cause Mortality (participants affected / at risk) | 0/634 | 0/900 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/634 | 0/900 | 0/19
Other Adverse Events (participants affected / at risk) | 0/634 | 0/900 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Hyperparathyroidism - Incomplete Data (N=634) | Primary Hyperparathyroidism (N=900) | DOTATATE and F-DOPA (N=19)
Abdominal pain (Gastrointestinal disorders) | NA | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT00001277/Prot_SAP_000.pdf